CLINICAL TRIAL: NCT02084810
Title: A Single Centre, Randomised, Double-blind, Two-way Crossover Trial in Healthy Male Subjects Investigating the Bioequivalence of Eptacog Alfa A 6 mg and NovoSeven®
Brief Title: Investigating the Bioequivalence of Eptacog Alfa A 6 mg and NovoSeven® in Healthy Male Subjects
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN7777-4087; 2013-003163-63 (EudraCT Number); U1111-1145-6620 (Other: WHO)
Record Dates: First submitted 2014-01-28; First posted 2014-03-12 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-03

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia A With Inhibitors; Haemophilia B; Haemophilia B With Inhibitors; Healthy
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VII

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NovoSeven® (Active Comparator)
  Interventions: Drug: activated recombinant human factor VII
- Eptacog alfa A 6 mg (Experimental)
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: activated recombinant human factor VII — All subjects will receive one i.v. (intravenous, into the vein) injection of 90μg/kg.
  Each subject will be allocated to two treatment periods separated by a wash-out period of a week.
  Arms: NovoSeven®
Drug: eptacog alfa (activated) — All subjects will receive one i.v. injection of 90μg/kg. Each subject will be allocated to two treatment periods separated by a wash-out period of a week.
  Arms: Eptacog alfa A 6 mg

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the bioequivalence of eptacog alfa A 6 mg and NovoSeven® in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male, age 18-55 years, both inclusive, at the time of signing informed consent
* Body Mass Index (BMI) 18.5-30 kg/m^2, both inclusive
* Good general health based on assessment of medical history, vital signs, physical examination, ECG (electrocardiogram), and laboratory data at screening, as judged by the investigator

Exclusion Criteria:

* Known history of thromboembolic event(s) or potential thromboembolic risk as judged by the investigator

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Area under the curve | After a single i.v. injection based on FVIIa activity assessments up to 36 hours post dose
Maximum concentration | After a single i.v. injection based on FVIIa activity assessments up to 36 hours post dose

SECONDARY OUTCOMES:
Frequency of adverse events (including serious adverse events) | Assessed up to 7 weeks following first trial product administration
Incidence of antibodies | Assessed up to 7 weeks following first trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com